CLINICAL TRIAL: NCT03401047
Title: Study to Assess Potential Impairments in Estradiol Augmentation of Gonadotropin Secretion in Polycystic Ovary Syndrome
Acronym: CRM009
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Christine Burt Solorzano, Dr., MD, Associate Professor of Pediatric Endocrinology, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19692
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Estradiol

STUDY DESIGN:
Intervention Model Description: This is a prospective interventional cohort study. Women with PCOS and controls will receive identical treatment (transdermal estradiol) and will be monitored using the same surveillance protocol. The study does not involve randomization, and it is not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transdermal Estradiol (Experimental): Subjects will undergo estradiol administration for up to 9 days. Transdermal estradiol patches will be applied each day by study staff during study days two through nine (patches deliver 0.1 mg/day for a total dose of up to 0.6 mg/day).
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Estradiol — Subjects will receive graded doses of transdermal estradiol patches for up to 7 days. Blood estradiol tests will be performed daily, and the number of estradiol patches used will be adjusted to maintain serum estradiol levels of 250-400 pg/ml. Estradiol is a natural hormone.
  Other Names: Vivelle

SUMMARY:
The purpose of this study is to determine if estradiol augmentation of luteinizing hormone (LH) secretion secretion (primary endpoint) and follicle-stimulating hormone (FSH) secretion (secondary endpoint) is reduced in adult women with polycystic ovary syndrome.

DETAILED DESCRIPTION:
This is a two-group controlled study to test the following hypothesis: compared to body mass index (BMI)-matched normal controls, women with polycystic ovary syndrome (PCOS) will demonstrate blunted LH responses to preovulatory estradiol concentrations. We will study both normally-cycling controls and women with PCOS. We aim to recruit BMI-matched pairs (PCOS vs. control within 2 kg/m2). To provoke a gonadotropin surge, subjects will receive graded transdermal estradiol dosing, and we will use a dose adjustment protocol to maintain serum estradiol levels of 250-400 pg/ml. To enhance reliability of estradiol delivery, transdermal estradiol patches will be placed/replaced daily by Clinical Research Unit (CRU) nurses, and abdominal sites will be rotated. All subjects will begin estradiol on menstrual cycle day 4. Starting 24 hours before E2 administration, all subjects will collect all urine output in 12-hour time blocks for later urinary LH and FSH analysis; this will continue until the end of the study. Additionally, subjects will have daily morning blood draws in the CRU for later hormone measurements. Transvaginal ovarian ultrasound will be performed on study day 6 -- near the time of expected surge initiation -- to document largest follicle sizes. We will measure serum estradiol daily and employ an estradiol dose-adjustment protocol to maintain target estradiol levels. We will also measure LH daily. The study will be stopped after either (a) serum LH increases to 5-fold higher than baseline and subsequently falls to within 200% of baseline, or (b) the subject has received estradiol for a full 7 days, whichever comes first. The primary endpoint will be estradiol-induced change in 24-hour urinary LH excretion, defined as 24-hour mean values immediately prior to estradiol administration vs. peak 24-hour mean values during estradiol administration. A comparison of 24-hour LH changes between healthy normal and PCOS groups will be conducted by way of a random-effects analysis of covariance (ANCOVA) model. The ANCOVA model will be specified so that each BMI-matched pair will represent an independent observational unit with respect to comparing 24-hour LH change between groups. With regard to hypothesis testing, we will test whether the component of variability in 24-hour LH change attributed to "Study Group" (healthy normal control vs. PCOS) is a significant component of the overall variability in 24-hour LH change. Variability in 24-hour LH change attributed to baseline disparities in LH will be accounted for by treating subject-specific baseline LH as a covariate in the ANCOVA model. If BMI matching is inadequate, we will also include BMI as a covariate in the model. If 11 women with PCOS and 11 controls complete study, we expect at least 80% power to detect a 33% difference in E2-induced augmentation of urinary LH excretion.

ELIGIBILITY:
Inclusion Criteria:

* PCOS group: post-pubertal (> 4 years post-menarche) adult woman aged 18-30 years with PCOS, defined as clinical and/or laboratory evidence of hyperandrogenism (hirsutism and/or elevated serum [calculated] free testosterone concentration) plus ovulatory dysfunction (irregular menses, fewer than 9 per year), but without evidence for other potential causes of hyperandrogenism and/or ovulatory dysfunction
* Control group: post-pubertal (> 4 years post-menarche) adult woman aged 18-30 years with regular menstrual periods (every 26-35 days) and no evidence of hyperandrogenism (i.e., no hirsutism, normal serum [calculated] free testosterone concentration)
* General good health (excepting overweight, obesity, PCOS, and adequately-treated hypothyroidism)
* Capable of and willing to provide informed consent
* Willing to strictly avoid pregnancy with use of reliable non-hormonal methods during the study period

Exclusion Criteria:

* Inability/incapacity to provide informed consent
* Males will be excluded (hyperandrogenism is unique to females)
* Age < 18 years (we do not propose to study children because we have no preliminary data that would support this particular study in children)
* Age > 30 years (since ovarian reserve may decrease beyond age 30)
* Obesity resulting from a well-defined endocrinopathy or genetic syndrome
* Positive pregnancy test or current lactation
* Evidence for non-physiologic or non-PCOS causes of hyperandrogenism and/or anovulation
* Evidence of virilization (e.g., rapidly progressive hirsutism, deepening of the voice, clitoromegaly)
* Total testosterone > 150 ng/dl, which suggests the possibility of virilizing ovarian or adrenal tumor
* DHEA-S greater than upper reference range limit for controls; and DHEA-S elevation > 1.5 times the upper reference range limit for PCOS. Mild elevations may be seen in PCOS, and will be accepted in this group.
* Early morning 17-hydroxyprogesterone > 200 ng/dl measured in the follicular phase, which suggests the possibility of congenital adrenal hyperplasia (if elevated during the luteal phase, the 17-hydroxyprogesterone will be repeated during the follicular phase). NOTE: If a 17-hydroxyprogesterone > 200 ng/dl is confirmed on repeat testing, an ACTH stimulated 17-hydroxyprogesterone < 1000 ng/dl will be required for study participation.
* Abnormal thyroid stimulating hormone (TSH): Note that subjects with stable and adequately treated primary hypothyroidism, reflected by normal TSH values, will not be excluded.
* Hyperprolactinemia: Any degree of hyperprolactinemia (confirmed on repeat) will be grounds for exclusion for subjects without PCOS. Hyperprolactinemia > 20% higher than the upper limit of normal will be grounds for exclusion for subjects without PCOS. Mild prolactin elevations may be seen in PCOS, and elevations within 20% higher than the upper limit of normal will be accepted in this group.
* History and/or physical exam findings suggestive of Cushing's syndrome, adrenal insufficiency, or acromegaly
* History and/or physical exam findings suggestive of hypogonadotropic hypogonadism (e.g., symptoms of estrogen deficiency) including functional hypothalamic amenorrhea (which may be suggested by a constellation of symptoms including restrictive eating patterns, excessive exercise, psychological stress, etc.)
* Persistent hematocrit < 36% and hemoglobin < 12 g/dl
* Severe thrombocytopenia (platelets < 50,000 cells/microliter) or leukopenia (total white blood count < 4,000 cells/microliter)
* Previous diagnosis of diabetes, fasting glucose > or = 126 mg/dl, or a hemoglobin A1c > or = 6.5%
* Persistent liver panel abnormalities, with two exceptions. Mild bilirubin elevations will be accepted in the setting of known Gilbert's syndrome. Also, mild transaminase elevations may be seen in obesity/PCOS; therefore, elevations < 1.5 times the upper limit of normal will be accepted in these groups.
* Significant history of cardiac or pulmonary dysfunction (e.g., known or suspected congestive heart failure, asthma requiring intermittent systemic corticosteroids, etc.)
* Decreased renal function evidenced by GFR < 60 ml/min/1.73m2
* A personal history of breast, ovarian, or endometrial cancer
* History of any other cancer diagnosis and/or treatment (with the exception of basal cell or squamous cell skin carcinoma) unless they have remained clinically disease free (based on appropriate surveillance) for five years
* History of allergy to transdermal estradiol patches
* BMI < 18 or > 40 kg/m2; BMI < 18 kg/m2 is considered to be underweight, while > 40 kg/m2 is considered to be class 3 obesity -- both may have marked confounding effects for the outcomes of interest
* Menstrual cycles lasting fewer than 26 days: Cycle frequency < 26 days suggest the possibility of relatively short follicular phases (e.g., < 12 days). If a subject with a follicular phase shorter than 12 days participates in Aim 1c, they could experience an endogenous gonadotropin surge under surveillance. Since we wish to capture only experimentally-induced surges, we will exclude such subjects.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Estimated)
Dates: Start 2017-11-30 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Estradiol-induced change in 24-hour urinary LH excretion | Change occurring over up to 7 days of estradiol administration
  The estradiol-induced change in 24-hour urinary LH excretion is defined as the 24-hour urinary LH excretion immediately prior to estradiol administration vs. the peak 24-hour urinary LH excretion during estradiol administration.

SECONDARY OUTCOMES:
Estradiol-induced change in 24-hour urinary FSH excretion | Change occurring over up to 7 days of estradiol administration
  The estradiol-induced change in 24-hour urinary FSH excretion is defined as the 24-hour urinary FSH excretion immediately prior to estradiol administration vs. the peak 24-hour urinary FSH excretion during estradiol administration.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Burt Solorzano, M.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Clinical Research Unit, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT03401047/Prot_SAP_000.pdf